CLINICAL TRIAL: NCT02700958
Title: Study of Remote Ischemic Preconditioning as a Preventative Method Against Subclinical Renal Injury and Contrast-induced Nephropathy
Brief Title: Remote Ischemic Preconditioning as a Method Against Subclinical Renal Injury and Contrast-induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tartu University Hospital (Other)
Responsible Party: Principal Investigator, Jaak Kals, Tartu University Hospital, Clinic of Surgery, Department of Vascular Surgery, cardiovascular surgeon; MD-PhD, Tartu University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16003
Record Dates: First submitted 2016-02-03; First posted 2016-03-07 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Atherosclerosis; Stable Angina; Peripheral Artery Disease; Contrast-induced Nephropathy
Keywords: Remote ischemic preconditioning; Contrast-induced Nephropathy; Stable coronary artery disease; Lower extremity arterial disease; Low molecular weight metabolites; Functional properties of arteries
MeSH Terms: conditions — Atherosclerosis; Angina, Stable; Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Remote ischemic preconditioning (Experimental): Remote Ischemic Preconditioning (RIPC) is performed by inflating blood pressure cuff for 5-minutes at 200 mmHg, or if patients systolic blood pressure is higher than 200 mmHg 20 mmHg above systolic pressure, alternated with 5-minute deflation for 4 times.
  Interventions: Procedure: Remote ischemic preconditioning
- SHAM remote ischemic preconditioning (Sham Comparator): SHAM Remote Ischemic Preconditioning (RIPC-SHAM) is accomplished by alternating 4 cycles of 5-minute inflation with 5-minute deflation. Blood pressure cuff will be inflated to 10-20 mmHg. RIPC-SHAM is performed with standard blood pressure cuff on upper-arm.
  Interventions: Procedure: SHAM Remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning is performed with standard blood pressure cuff on upper-arm. RIPC will be started just before the coronarography or angiography. Time between the last inflation cycle and the beginning of the procedure will be less than 60 minutes.
  Arms: Remote ischemic preconditioning
Procedure: SHAM Remote ischemic preconditioning — SHAM Remote ischemic preconditioning is performed with standard blood pressure cuff on upper-arm. RIPC-SHAM will be started just before the coronarography or angiography. Time between the last inflation cycle and the beginning of the procedure will be less than 60 minutes
  Arms: SHAM remote ischemic preconditioning

SUMMARY:
Contrast-induced nephropathy (CIN) has remained significant and severe complication of angiographic procedures despite the increasing use of preventative methods. It has been associated with prolonged hospital stay, high morality and the need for dialysis. Since classically used creatinine for diagnosing of CIN does not reflect the degree of tubular injury before 24-48 hours after exposure to contrast media alternative earlier biomarkers and preventative methods are needed. Remote ischemic preconditioning is a non-invasive and safe method which in some studies has been reported to protect against contrast-induced nephropathy. The purpose of this study is to evaluate the effect of remote ischemic preconditioning (RIPC) (1) as an additional method to standard treatment to prevent subclinical and clinical contrast-induced acute kidney injury and (2) to assess its effect on functional properties of arterial wall, organ damage biomarkers and low molecular weight metabolites.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years, no upper age limit
* Patients with stable coronary artery disease (II - III class according to the Canadian Cardiovascular Society) hospitalized for coronarography or with lower extremity arterial disease hospitalized for angiography
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Age less than 18 years
* eGFR < 30 ml/min/1,73 m2
* Simultaneous participation in an other clinical trial
* Coexisting pathology of the upper-limbs limiting the use of the cuff (bilateral amputee, recent trauma, chronic ulcers, significant upper limb peripheral atherosclerosis (radial pulse not palpable on either side))
* Malignant tumor (in remission less than 5 years or ongoing treatment)
* Documented allergic reaction to iodinated contrast agent
* Acute infection (body temperature 38 degrees Celsius or higher, c reactive protein 50mg/L or higher)
* Cardiac rhythm abnormalities (atrial fibrillation, frequent supraventricular premature complexes)
* Documented myocardial infarction within 30 days
* Inability to understand the instructions of the study
* Vascular surgery in axillary region
* Unable to lie supine for 40 minutes
* Home oxygen treatment
* Documented upper limb deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2019-03-19

PRIMARY OUTCOMES:
Change in carotid-femoral pulse wave velocity compared with baseline and SHAM subgroup | 24 hours
  Carotid-femoral pulse wave velocity baseline measurement is performed. Second measuring is performed 24 hours after angiographic procedure. Change from baseline will be compared between RIPC and SHAM subgroups. Measuring is performed with SphygmoCor XCEL PWA and PWV Device.
Change in augmentation indices (augmentation index and heart rate-corrected augmentation index (AIx@75)) compared with baseline and SHAM subgroup | 24 hours
  Augmentation indices baseline measurement is performed. Second measuring is performed 24 hours after angiographic procedure. Change from baseline will be compared between RIPC and SHAM subgroups. Measuring is performed with SphygmoCor XCEL PWA and PWV Device.

SECONDARY OUTCOMES:
Cardiac markers | 24 hours
  N-terminal pro-brain natriuretic peptide (NT-proBNP), creatine kinase (CK) MB isoenzyme, troponin T
Traditional biomarkers of renal function | 24 hours
  Urea, creatinine
Novel biomarkers of renal function | 24 hours
  Neutrophil gelatinase-associated lipocalin (NGAL), renal liver-type fatty acid binding protein (L-FABP), kidney injury molecule-1 (KIM-1), isoprostane, cystatin C, beta-2 microglobulin
Estimated glomerular filtration rate | 24 hours
  eGFR
Markers of oxidative stress and inflammation | 24 hours
  Oxidized low density lipoprotein (oxLDL), interleukin 18 (IL-18), myeloperoxidase (MPO)
Length of hospital stay | 30 days
  Length of hospital stay measured in days.
Adverse events of angiographic procedures | 7 days
  Allergic reactions to iodinated contrast media or local anesthetics
All-cause and cardiovascular mortality | 1 year
  Data of 1-year all-cause and cardiovascular mortality will be collected from the Estonian Causes of Death Registry.
Adverse events associated with femoral artery puncture | 24 hours
  Bleeding, hematoma, arterial thrombosis
Cardiac event | 30 days
  Myocardial infarction or cardiac arrest
Adverse events of remote ischemic preconditioning | 10 days
  Upper-extremity deep vein thrombosis, acute upper limb ischaemia
Low molecular weight metabolites | 24 hours
  Amino acids (alanine, arginine, asparagine, aspartate, citrulline, cysteine, glutamine, glutamate, glycine, histidine, hydroxyproline, leucine, lysine, methionine, ornithine, phenylalanine, proline, serine, threonine, tryptophan, tyrosine, valine), acylcarnitines (free carnitine, acylcarnitine, propionylcarnitine, butyrylcarnitine, pentanoylcarnitine, hexanoylcarnitine, octanoylcarnitine, decanoylcarnitine, tetradecanoylcarnitine, octadecanoylcarnitine), hydroxy acids and other metabolic parameters (aconitate, α-ketoglutarate, β-hydroxybutyrate, citrate, citrulline, 7-ketocholesterol, lactate, malonate, oxaloacetate, pyruvate, succinate) will be measured.
Arterial elasticity indices | 24 hours
  Arterial elasticity indices baseline measurement is performed. Second measuring is performed 24 hours after angiographic procedure. Change from baseline will be compared between RIPC and SHAM subgroups. Measuring is performed with HD/PulseWave™ CR-2000.

CONTACTS AND LOCATIONS:
Overall Officials: Jaan Eha, MD, PhD, Study Chair — Tartu University Hospital; Jaak Kals, MD, PhD, Principal Investigator — Tartu University Hospital; Mihkel Zilmer, MD, PhD, Study Chair — University of Tartu; Karl Kuusik, MD, Study Director — University of Tartu; Teele Kepler, MD, Study Chair — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Tartu County, Estonia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liang F, Liu S, Liu G, Liu H, Wang Q, Song B, Yao L. Remote ischaemic preconditioning versus no remote ischaemic preconditioning for vascular and endovascular surgical procedures. Cochrane Database Syst Rev. 2023 Jan 16;1(1):CD008472. doi: 10.1002/14651858.CD008472.pub3. PMID 36645250